CLINICAL TRIAL: NCT04054284
Title: Safety and Efficacy of a Complex Herbal Tea Mixture in Type 2 Diabetics
Brief Title: Safety and Efficacy of Herbal Tea in Type 2 Diabetics
Acronym: DIABHerbMix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Collaborators: Dom zdravlja Osijek (Health Centre Osijek) (Unknown); Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Ines Banjari, Associate Prof. Dr., Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: JJStrossmayerU-1
Record Dates: First submitted 2019-07-29; First posted 2019-08-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes; Herbal Medicine Adverse Reaction
Keywords: Type 2 Diabetes; Herbal Medicine; Safety; Glycaemia Control; Alternative Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Teas, Herbal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Herbal Tea Mixture is consisted of: Vaccinium myrtillus L. folium, Morus nigra L. folium, Phaseolus vulgaris L. pericarpium, Viscum album L. herba, Urtica dioica L. radix, Gentiana lutea L. radix, Taraxacum officinale W. radix, Cichorium intybus L. herba, Teucrium chamaedrys L. herba, Stevia rebaudiana folium.
  Interventions: Dietary Supplement: Antidiabetic Herbal Tea
- Control (Active Comparator): Herbal Tea Mixture without antidiabetic properties is consisted of: Achillea millefolium L. herba, Teucrium montanum L. herba, Glechoma hederacea L. herba, Eupatorium cannabinum L. herba, Humulus lupulus L. lupulin, Artemisia absinthium L. herba, Salvia officinalis L.
  Interventions: Dietary Supplement: Herbal Tea

INTERVENTIONS:
Dietary Supplement: Antidiabetic Herbal Tea — Patients will be instructed to take 250 mL of freshly prepared tea (1 tea spoon or 3 g of tea, pour over 250 mL of boiling water and leave aside for 15 min) 2 times per day during 12 weeks. The first tea needs to be taken in the morning prior any meal. The second can be taken at any time during the day but with at least 4 hour difference from the first cup.
  Other Names: Experimental-Intervention
  Arms: Intervention
Dietary Supplement: Herbal Tea — Patients will be instructed to take 250 mL of freshly prepared tea (1 tea spoon or 3 g of tea, pour over 250 mL of boiling water and leave aside for 15 min) 2 times per day during 12 weeks. The first tea needs to be taken in the morning prior any meal. The second can be taken at any time during the day but with at least 4 hour difference from the first cup.
  Other Names: Active Comparator-Control
  Arms: Control

SUMMARY:
Nearly 25% of the world's population relies on traditional medicinal systems but for professionals their effectiveness and even more safety are the main concern. Therefore, the aim of this preliminary study is to assess safety and effectiveness of herbal tea mixture on the control of glycaemia in Type 2 diabetics.The mixture consists of nine plants which have well-documented traditional use for the control of glycaemia.

DETAILED DESCRIPTION:
The study will include Type 2 Diabetics who are taking only oral hypoglycemic medications (without insulin). Their therapy has to be stable for at least 3 months prior enrollment. Besides anthropometric measures, patient's glycaemia, renal and liver function will be monitored. Safety and adverse events will be closely monitored and these are the primary outcomes of the study. The main outcome measure of the effectiveness is HbA1c (glycated hemoglobin). Patients will be given detailed instructions on how to prepare the tea and the dosing. The intervention will last 3 months and during that time patients will be asked not to change their dietary or lifestyle habits.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* Croatian-speaking
* stable therapy for at least 3 months prior enrollment
* not taking any dietary supplements, especially herbal-based
* not taking any other herbal medicine (as a tea or a supplement)
* stable dietary and lifestyle patterns for at least 3 months prior enrollment

Exclusion Criteria:

* type 1 diabetes
* severe somatic disorder (oncological disease, hepatic, renal or autoimmune disease)
* pregnancy
* inability to fill in questionnaires in Croatian
* cognitive impairment
* psychiatric disorder
* undergoing current treatment for a major medical illness such as malignancy, autoimmune or immune deficiency disorder
* clotting disorders
* having nutritional deficiency (e.g. iron deficiency)
* current or history of eating disorder (anorexia, bulimia or EDNOS)
* current use of weight loss interventions (drugs; exercise interventions)
* regular use of dietary supplements, especially herbal-based
* regular use of herbal medicine (as a tea or a supplement)
* significant changes in diet or lifestyle patterns (e.g. increased physical activity) in the last 3 months prior the enrollment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse event | Starting from baseline, once per week until study completion at week 12.
  Adverse event (e.g. hypoglycaemia) reporting through direct contact researcher-patient.

SECONDARY OUTCOMES:
Glycated Hemoglobin | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood HbA1c (%)
Fasting Glucose | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood Glucose (mmol/L)

OTHER OUTCOMES:
Creatinine | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of Creatinine (µmol)
Urea | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of Urea (mmol/L)
Total Proteins | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of Total Proteins (g/L)
Alanine transaminase | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of liver enzymes Alanine transaminase (ALT in U/L)
Aspartate transaminase | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of liver enzymes Aspartate transaminase (AST in U/L)
Alkaline phosphatase | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of liver enzymes Alkaline phosphatase (ALP in U/L)
Gamma-glutamyl transpeptidase | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Blood concentration of liver enzymes Gamma-glutamyl transpeptidase (GGT in U/L)
Body Weight | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Change in body weigh (in kg), Body Mass Index in kg/m2, waist circumference in cm
Body Mass Index | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Change in Body Mass Index (kg per square meter)
Waist Circumference | At enrollment (baseline) and at the end of the intervention (at 12 weeks).
  Change in waist circumference (in cm)

CONTACTS AND LOCATIONS:
Overall Officials: Ines Banjari, PhD, Principal Investigator — Department of Food and Nutrition Research, Faculty of Food Technology
Locations (3):
- Croatia (3):
  - Department of Food and Nutrition Research, Faculty of Food Technology, Osijek
  - Health Centre Osijek, Osijek
  - University Hospital Centre, Osijek